CLINICAL TRIAL: NCT03666234
Title: Idiopathic Pulmonary Fibrosis Registry China Study
Acronym: PORTRAY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dai Huaping (Other)
Responsible Party: Sponsor-Investigator, Dai Huaping, Deputy Director of Center for Respiratory Diseases, China-Japan Friendship Hospital
Organization: China-Japan Friendship Hospital (Other)
Other Study IDs: ChinaJapanFH002
Record Dates: First submitted 2018-06-20; First posted 2018-09-11 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic Pulmonary Fibrosis; Epidemiology; Nature History
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
By mean of registry of newly diagnosed Chinese IPF patients from more than 15 sites, this study aims to build IPF prospective cohort, set up normative clinical database and a biological specimen bank, and examine the clinical characteristics of newly diagnosed Chinese IPF patients, as well as the nature history, prognosis, comorbidities and complications of IPF patients in China, the current treatment pattern, burden of illness, and quality of life of Chinese IPF patients.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosed IPF during the last 3 months based upon ATS/ERS/JRS/ALAT guidelines 2011
* Aged 40 years and above at recruitment
* Willing and able to sign an informed consent

Exclusion Criteria:

* Inclusion in any interventional clinical trials
* Lung transplantation expected within the next 6 months.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chinese newly diagnosed IPF patients
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Demographic and clinical characteristic of newly diagnosed Chinese IPF patients | up to 5 years
  Data analyses will be mainly descriptive.

SECONDARY OUTCOMES:
Mortality in Chinese patients with IPF | up to 5 years
  Mortality will be showed as percentage.
Cause of death in Chinese patients with IPF | up to 5 years
  Cause of death:
  a. IPF-related: i. Respiratory failure: Pulmonary failure leads to impaired gas exchange, i.e. hypoxemia and/or hypercapnia ii. Acute exacerbation of IPF (as defined below) iii. Other aspects related to IPF (please specify); b. Concomitant conditions: i. Coronary heart disease ii. Cerebrovascular disease iii. Pneumonia/respiratory tract infection iv. Pulmonary embolism v. Pulmonary hypertension or pulmonary hypertension/right heart failure vi. Lung cancer; c. Other causes; d. Unknown.
  Cause of death will be showed as categorical variable, and the counts and percentile ratios will be statistically counted.
Progression-free survival in Chinese patients with IPF | up to 5 years
  Patients without the following events:
  1. Death
  2. Lung transplantation
  3. Acute exacerbation
  4. Require long-term oxygen therapy
  5. Hospitalization for respiratory reasons
  The unit of progression-free survival is day.
Description of the acute exacerbations in Chinese patients with IPF | up to 5 years
  Acute exacerbation of IPF (AE-IPF)
  1. Previous diagnosis or simultaneous diagnosis of IPF;
  2. Symptoms generally manifest as dyspnea with acute exacerbations or progression within 1 month;
  3. Chest CT shows new bilateral glass ground or solid shadows on the basis of usual interstitial pneumonia (UIP);
  4. Exacerbations cannot be completely explained by heart failure or increased volume load.
  The incidence of the acute exacerbation will be showed as percentage.

CONTACTS AND LOCATIONS:
Locations (1):
- Huaping Dai, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang X, Wang H, Liu A, Ni Y, Wang J, Han Y, Xie B, Geng J, Ren Y, Zhang R, Liu M, Dai H. Evaluation of respiratory muscle dysfunction in patients with idiopathic pulmonary fibrosis: a prospective observational study with magnetic resonance imaging. BMC Pulm Med. 2025 Mar 14;25(1):118. doi: 10.1186/s12890-025-03572-6. PMID 40087606
- [Derived] Xie B, Ren Y, Geng J, He X, Ban C, Wang S, Jiang D, Luo S, Chen Q, Liu M, Feng R, Zhao L, Dai H, Wang C. Idiopathic Pulmonary Fibrosis Registry China study (PORTRAY): protocol for a prospective, multicentre registry study. BMJ Open. 2020 Nov 11;10(11):e036809. doi: 10.1136/bmjopen-2020-036809. PMID 33177132